CLINICAL TRIAL: NCT05699811
Title: Phase I/II Trial of Allograft Engineered MSC-IFNα Combined With or Without Immunochemotherapy for Locally Advanced/Metastatic Solid Tumors
Brief Title: IFNα Expressing Mesenchymal Stromal Cells for Locally Advanced/Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Collaborators: Wuxi Sinotide New Drug Discovery Institutes (Unknown)
Responsible Party: Principal Investigator, Han weidong, Director of Biotherapeutic Department, Chinese PLA General Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-078
Record Dates: First submitted 2023-01-07; First posted 2023-01-26 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Locally Advanced or Metastatic Solid Tumors
MeSH Terms: interventions — Taxes; Albumin-Bound Paclitaxel; Cyclophosphamide; spartalizumab; toripalimab; sintilimab; camrelizumab; tislelizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MSC-IFNα monotherapy (Experimental): Subjects will be enrolled for safety evaluation of MSC-IFNα monotherapy. Subjects will receive MSC-IFNα infusion from a dose of 2×10^6 cells/kg 1-4 times every 4-6 weeks. All treatment-related adverse events(TRAE) will be recorded for at least 28 days after the cell infusion.
  Interventions: Biological: MSC-IFNα
- MSC-IFNα combined with immunochemotherapy (Experimental): Subjects will be enrolled and received MSC-IFNα combined with immunochemotherapy, namely nab-paclitaxel (125 mg/m2, 5 days before infusion), cyclophosphamide (200 mg/m2,4 days before infusion) and anti-PD-1 antibody (200mg, 7 days after infusion) for 4 cycles.
  From the 5th cycle, subjects will receive MSC-IFNα combined with anti-PD-1 antibody every 4-6 weeks for another 4 cycles for efficacy consolation. From the 9th cycle, subjects will receive anti-PD-1 antibody alone every 3 weeks for another 4 cycles for efficacy maintenance.
  Interventions: Biological: MSC-IFNα; Drug: Nab paclitaxel; Drug: Cyclophosphamide; Drug: Anti-PD-1 monoclonal antibody

INTERVENTIONS:
Biological: MSC-IFNα — MSC-IFNα form a dose of 2×10^6 cells/kg, intravenous infusion every 4-6 weeks
Drug: Nab paclitaxel — 125mg/m2, intravenous infusion every 4-6 weeks
  Other Names: Abraxane
  Arms: MSC-IFNα combined with immunochemotherapy
Drug: Cyclophosphamide — 200mg/m2, intravenous infusion every 4-6 weeks
  Arms: MSC-IFNα combined with immunochemotherapy
Drug: Anti-PD-1 monoclonal antibody — 200mg, intravenous infusion every 4-6 weeks
  Other Names: Toripalimab Injection; Sintilimab Injection; Camrelizumab Injection; Tislelizumab Injection
  Arms: MSC-IFNα combined with immunochemotherapy

SUMMARY:
The goal of this first-in-human, single-center, prospective, open-label, phase 1/2 trial is to evaluate the safety and efficacy of the interferon alpha expressing mesenchymal stromal cells (MSC-IFNα) combined with or without immunochemotherapy in patients with locally advanced/metastatic solid tumors. The main questions aimed to answer are 1) to evaluate the safety and feasibility of MSC-IFNα in the treatment of locally advanced/metastatic solid tumors;2) to evaluate the anti-tumor effects of the MSC-IFNα combined with or without immunochemotherapy in the treatment of locally advanced/metastatic solid tumors; 3) to evaluate the pharmacokinetics/pharmacodynamics of MSC-IFNα and related immune effector cells.

DETAILED DESCRIPTION:
[Introduction] Mesenchymal Stromal Cells (MSCs) have been shown to home to the sites of injury or damage and secrete immunomodulatory factors. This feature makes MSCs an ideal carrier to deliver drugs or cytokines to the tumor microenvironment (TME) and therefore have a potential therapeutic role in cancer treatment.

Interferon(IFN) has been widely used for cancer treatment for its pleiotropic antitumor effects. IFN receptor signals mediate intrinsic and extrinsic effects on tumor cells and the TME, including tumor-infiltrating lymphocytes as well as tumor-associated stroma. Additionally, IFNs also exert direct intrinsic antitumor effects including inhibition of cell proliferation by inducing cell cycle arrest, cell death via apoptosis and ferroptosis, cell differentiation, and senescence, thus acting as a tumor suppressor. Accumulating evidence suggests that IFNs play critical roles in cancer immunotherapy, however, the variations in responses and the adverse effects have reduced their popularity in clinical applications. New IFN-based strategies should be considered as a high priority.

Our team has developed a protocol to genetically express IFNα in bone marrow-derived MSCs. In vitro and in vivo experiments have shown that the MSC-IFNα cells possess a potent ability to home to TME and to secret IFNα. By changing TME, MSC-IFNα induces strong anti-tumor effects in several cancer types in animal models. In addition, preliminary data also indicated that the combination of IFNα-MSCs with chemotherapy and/or programmed death-1(PD-1)/programmed death-ligand 1(PD-L1)blockade may bring an even stronger anti-tumor immunity.

In this study, by producing MSC-IFNα cells with human umbilical-cord-derived mesenchymal stromal cells (hUC-MSCs, passage 5 to passage 7), the investigators plan to conduct a first-in-human, prospective, open-label, phase 1/2 trial to evaluate the safety and efficacy of MSC-IFNα combined with or without immunochemotherapy in patients with locally advanced/metastatic solid tumors.

[Study design] Phase 1 Arm 1. Safety evaluation of MSC-IFNα monotherapy A total of 3-9 subjects will be enrolled for the safety evaluation of MSC-IFNα monotherapy. All treatment-related adverse events (TRAE) will be recorded for at least 28 days after cell infusion. Subjects with any grade 3-4 TRAE that lasts for 7 days or more within the 28 days after infusion will be determined as treatment intolerance (TI).

The first 3 subjects will receive MSC-IFNα infusion 1-4 times every 4-6 weeks at a dose of 2×10^6 cells/kg. If TI occurred in any of the 3 subjects, another 3 subjects will be enrolled and received a 70% reduced MSC-IFNα dose (i.e. 6×10^5 cells/kg, 2x10^5/kg, and so on) until tolerable dose (no TI in all 3 subjects) was reached.

Arm 2. Safety and efficacy evaluation of MSC-IFNα combined with immunochemotherapy.

A total of 3-9 subjects will be enrolled and receive MSC-IFNα infusion (tolerable dose determined in Arm 1) every 4-6 weeks for 4 cycles. Immunochemotherapy, namely nab-paclitaxel (125 mg/m2, 5 days before cell infusions), cyclophosphamide (200 mg/m2,4 days before cell infusions) and anti-PD-1 antibody (200mg, 7 days after infusion) will be given. From the 5th cycle, subjects will receive MSC-IFNα combined with anti-PD-1 antibody (200mg, 7 days after infusion) every 4-6 weeks for another 4 cycles for efficacy consolation. From the 9th cycle, subjects will receive anti-PD-1 antibody (200mg) alone every 3 weeks for another 4 cycles for efficacy maintenance. The safety, efficacy, and other required data will be collected and the optimized combined regimen (OCR) of MSC-IFNα and immunochemotherapy will be determined. MSC-IFNα related AE will be continuously monitored in this arm, and reduced MSC-IFNα dose will be considered if necessary.

Phase 2 A total of 10-30 subjects will be enrolled and received the OCR determined in the phase 1 of the trial. The safety, efficacy, and other required data will be collected.

During the treatment, efficacy in all subjects will be assessed at baseline and every 8 weeks thereafter until confirmed progressive disease, death, intolerable toxicity, withdrawal of consent, or end of the study, whichever occurs first.

During post-treatment follow-up, efficacy and TRAEs in all subjects will be assessed every 12 weeks until death, withdrawal of consent, loss to follow-up, or end of the study, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 75 years with estimated life expectancy >3 months.
2. Histopathological confirmed locally advanced or metastatic solid tumors including, but not limited to, lung cancer, breast cancer, colorectal cancer, hepatocellular carcinoma, and sarcomas.
3. Failed to at least first-line and second-line treatments or initially diagnosed locally advanced/metastatic solid tumors that have no National Comprehensive Cancer Network(NCCN) guideline-recommended therapy.
4. Have at least one measurable target lesion.
5. Previous treatment must be completed for more than 4 weeks prior to the enrollment of this study.
6. Have an Eastern Cooperative Oncology Group performance status (ECOG) of 0 to 2 at the time of enrollment.
7. Have adequate organ function, which should be confirmed within 2 weeks prior to the first dose of study drugs.
8. Previous treatment with anti-PD-1/PD-L1 antibodies is allowed.
9. Ability to understand and sign a written informed consent document.
10. Women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and up to 90 days after the last dose of the drug.

Exclusion Criteria:

1. Active, known, or suspected autoimmune diseases.
2. Known brain metastases or active central nervous system (CNS). Subjects with CNS metastases who were treated with radiotherapy for at least 3 months prior to enrollment, have no central nervous symptoms, and are off corticosteroids, are eligible for enrollment, but require a brain MRI screening.
3. Subjects are being treated with either corticosteroid (>10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of enrollment.
4. History of psychiatric disorders including depression, suicidality, and mania.
5. History of allergy or intolerance to study drug components.
6. Substance abuse, medical, psychological, or social conditions that may interfere with the patient's participation in the study or evaluation of the study results.
7. Uncontrolled concurrent illness, including ongoing or active systemic infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia (excluding insignificant sinus bradycardia and sinus tachycardia), or psychiatric illness/social situations and any other illness that would limit compliance with study requirements and jeopardize the safety of the patient.
8. History of human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS).
9. Pregnant or breast-feeding. Women of childbearing potential must have a pregnancy test performed within 7 days before enrollment, and a negative result must be documented.
10. Previous or concurrent cancer within 3 years prior to treatment start.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-02-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment related adverse events(TRAE) | Up to 12 months since the initiation of MSC-IFNα therapy
  Treatment related adverse events (TRAE) are defined as any medical events since the initiation of MSC-IFNα therapy. All TRAEs will be recorded and graded according to the Common Terminology Criteria for Adverse Events (CTCAE V5.0)

SECONDARY OUTCOMES:
Objective response rate (ORR) of MSC-IFNα combined with or without immunochemotherapy | Up to 12 months since the initiation of MSC-IFNα therapy
  Objective response rate (ORR) is defined as the proportion of patients with a complete response or partial response to MSC-IFNα treatment according to Response Evaluation Criteria in Solid Tumors (RECIST 1.1) or immune RECIST (iRECIST)
Progression free survival (PFS) of MSC-IFNα combined with or without immunochemotherapy | Up to 12 months since the initiation of MSC-IFNα therapy
  Progression free survival (PFS) is defined as the time from enrollment of the study to disease progression or death from any cause.
Duration of response(DOR) of MSC-IFNα combined with or without immunochemotherapy | Up to 12 months since the initiation of MSC-IFNα therapy
  Duration of response(DOR) is defined as the length of time that a tumor continues to respond to treatment without the cancer growing or spreading
Overall survival (OS) of MSC-IFNα combined with or without immunochemotherapy | Up to 12 months since the initiation of MSC-IFNα therapy
  Overall survival (OS) is defined as the time from treatment to death, regardless of disease recurrence

OTHER OUTCOMES:
Allograft MSC-IFNa cells in peripheral blood and in tumor microenvironments. | Up to 12 months since the initiation of MSC-IFNα therapy
  Engineered MSC-IFNa will be periodically monitored by quantitative polymerase chain reaction (qPCR)
Serum interferon-α level after infusion of MSC-IFNα | Up to 12 months since the initiation of MSC-IFNα therapy
  Serum interferon-α level will be dynamically monitored by enzyme-linked immunosorbent assay (ELISA)
Serum interferon-β level after infusion of MSC-IFNα | Up to 12 months since the initiation of MSC-IFNα therapy
  Serum interferon-β level will be dynamically monitored by enzyme-linked immunosorbent assay (ELISA)
Serum interleukin-2 level after infusion of MSC-IFNα | Up to 12 months since the initiation of MSC-IFNα therapy
  Serum interleukin-2 level will be dynamically monitored by enzyme-linked immunosorbent assay (ELISA)
Serum interleukin-6 level after infusion of MSC-IFNα | Up to 12 months since the initiation of MSC-IFNα therapy
  Serum interleukin-6 level will be dynamically monitored by enzyme-linked immunosorbent assay (ELISA)
Serum tumor necrosis factor-α level after infusion of MSC-IFNα | Up to 12 months since the initiation of MSC-IFNα therapy
  Serum tumor necrosis factor-α level will be dynamically monitored by enzyme-linked immunosorbent assay (ELISA)
Dynamic changes of monocytes in peripheral blood after infusion of MSC-IFNα | Up to 12 months since the initiation of MSC-IFNα therapy
  Dynamic changes of monocytes (CD14+/CD16+) cell number and proportion in peripheral blood will be monitored by flow cytometry
Dynamic changes of CD4 T cells in peripheral blood after infusion of MSC-IFNα | Up to 12 months since the initiation of MSC-IFNα therapy
  Dynamic changes of CD4 T cells (CD3+/CD4+) cell number and proportion in peripheral blood will be monitored by flow cytometry
Dynamic changes of CD8 T cells in peripheral blood after infusion of MSC-IFNα | Up to 12 months since the initiation of MSC-IFNα therapy
  Dynamic changes of CD8 T cells (CD3+/CD8+) cell number and proportion in peripheral blood will be monitored by flow cytometry
Dynamic changes of nature killer (NK) cells in peripheral blood after infusion of MSC-IFNα | Up to 12 months since the initiation of MSC-IFNα therapy
  Dynamic changes of nature killer (NK) cells (CD3-/CD16+/CD56+) cell number and proportion in peripheral blood will be monitored by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: WeiDong Han, PhD, Principal Investigator — Chinsese PLA Gereral Hospital; Yufang Shi, PhD, Study Chair — Wuxi Sinotide New Drug Discovery Institutes
Locations (1):
- Department of Biotherapeutic, Chinese PLA General Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: In vitro and in vivo studies of MSC-IFN-α — https://www.nature.com/articles/s41388-022-02201-4